CLINICAL TRIAL: NCT02390661
Title: Drain Placement for Seroma Prevention After Mammosite/SAVI Catheter Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Harvey Bumpers, Professor of Surgery, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-931M; i044456
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Infected Seroma After Surgical Procedure
Keywords: seroma; accelerated partial breast irradiation (APBI); breast lumpectomy; breast cancer
MeSH Terms: conditions — Seroma; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No drain (No Intervention): Control group
- Penrose drain placement (Experimental): Placement of a penrose drain after irradiation catheter is removed
  Interventions: Device: Penrose drain placement

INTERVENTIONS:
Device: Penrose drain placement — A penrose drain will be placed in the lumpectomy cavity after removal of the irradiation catheter
  Arms: Penrose drain placement

SUMMARY:
The proposed study is randomised controlled trial where informed and consenting patients who have a Mammosite/SAVI device placed, are randomized into two groups: a control group that has the device removed in the traditional manner without having a drain placed, and an experimental group that will have a penrose drain placed under sterile conditions at the time of removal of their device. The drain will be placed in the same site used for the APBI device and no additional surgery will be performed. The drain will remain for 2-3 days and it will be removed by the patient at home. They will return for their routine follow-up appointments and be monitored for development of a seroma with the use of standard ultrasound and physical exam. Hypothesis: Based on the null hypothesis there will be no difference in the rate of seroma formation after the APBI device removal if a drain is placed.

DETAILED DESCRIPTION:
The proposed study is randomised controlled trial where informed and consenting patients who have an APBI device placed, are randomized into two groups: a control group that has the device removed in the traditional manner without having a drain placed, and a experimental group that would have a penrose drain placed under sterile conditions at the time of removal of their device. The procedure will be performed at the MSU Surgery outpatient clinic by residents, the senior investigator or a trained nurse/PA. Additional data will be collected on each patient from their medical record including demographic data, cancer diagnosis, lesion size, date of procedure, date Mammosite/SAVI was inserted and removed, total dose of radiation, ER, PR, HER2Neu status, and any chemotherapy or hormone therapy being administered. Drains will remain in place for 2-3 days and will be removed by the patient upon removing the dressing. Patients will continue their antibiotic regimen prescribed while the APBI device was in place for the 2-3 days the drain is in place for infection prophylaxis. Patients will be followed for 4 weeks to determine if a seroma or other complication has developed. Patients in both the experimental and control groups will have the same standard follow up and monitoring for seroma development with the use of ultrasound. All postop cancer care will be standard and this study will not alter or delay any aspect of breast cancer treatment. Statistics will be performed and reported based upon data collected.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast cancer
* received accelerated partial breast irradiation

Exclusion Criteria:

* any metastatic breast cancer
* infection
* skin with radiation injury

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Development of lumpectomy cavity seroma | 1 month and 4 months
  The patient will be evaluated by physical exam and ultrasound of the affected breast.

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Bumpers, MD, Principal Investigator — Michigan State University, CHM
Locations (1):
- Michigan State University Dept Surgery/Sparrow Hospital, Lansing, Michigan, United States